CLINICAL TRIAL: NCT00482989
Title: A Phase 1b, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety and Tolerability of Multiple Intravenous Doses of MEDI-545, a Fully Human Anti-Interferon-Alpha Monoclonal Antibody, in Patients With Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Safety and Tolerability of Multiple Intravenous Doses of MEDI 545 in Patients With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP152; NCT00566163 (obsolete NCT alias)
Record Dates: First submitted 2007-06-04; First posted 2007-06-06 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Lupus
MeSH Terms: interventions — sifalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): MEDI-545
  Interventions: Biological: MEDI 545
- 2 (Other): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MEDI 545 — MEDI-545 is supplied as a sterile liquid containing 0.75 mL of MEDI-545 solution at a concentration of 100 mg/mL in a 3 mL single-use glass vial.
  Dosage, frequency and duration: MEDI-545 (0.3, 1.0, 3.0, or 10.0 mg/kg) will be administered via infusion over at least 60 minutes every 2 weeks for 26 weeks.
  Arms: 1
Other: Placebo — Dosage form: Placebo is supplied as a sterile liquid containing a 0.75 mL solution in a 3 mL single-use vial.
  Dosage, frequency and duration: Placebo (0.3, 1.0, 3.0, or 10.0 mg/kg) will be administered via infusion over at least 60 minutes every 2 weeks for 26 weeks.
  Arms: 2

SUMMARY:
To evaluate the safety and tolerability of multiple IV doses of the MEDIMUNNE antibody in adult patients with SLE.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of multiple IV doses of MEDI-545 in adult patients with SLE.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ≥ 18 years of age at the time of the first dose of study drug;
* Written informed consent obtained from the patient; or patient's legal representative;
* Meet at least 4 of the 11 revised ACR classification criteria for SLE (see Appendix A) (ACR,1999);
* Have positive ANA test at ≥ 1:80 serum dilution in the past or at screening;
* Have at least one system with a score of A or two systems with a score of B on the BILAG index at screening, or have a SELENA-SLEDAI score ≥ 6;
* Sexually active women, unless surgically sterile (including tubal ligation) or at least 2 years post-menopausal, must use an effective method of avoiding pregnancy (including oral, injectable, transdermal, or implanted contraceptives, intrauterine device, diaphragm with spermicide, cervical cap, abstinence, sterile sexual partner) in addition to the use of condoms (male or female condoms with spermicide) from screening through the end of the study. Cessation of birth control after this point should be discussed with a responsible physician. Sexually active men, unless surgically sterile, must likewise practice two effective methods of birth control (condom with spermicide or abstinence) and must use such precautions from Study Day 0 through the end of the study.
* Ability to complete the study period, including follow-up period through Study Day 350; and
* Willing to forego other forms of experimental treatment during study.

Exclusion Criteria:

* Have received MEDI-545 within 120 days prior to screening or have either detectable levels of MEDI-545 or anti-MEDI-545 antibodies (positive at > 1:10 serum dilution) in serum at screening;
* History of allergy or reaction to any component of the study drug formulation;
* Have received prednisone > 20 mg/day (or an equivalent dose of another oral corticosteroid)within 14 days before randomization/entry;
* Have received the following dosages of medications within 28 days before randomization/entry: hydroxychloroquine > 600 mg/day, mycophenolate mofetil > 3 g/day,methotrexate > 25 mg/week, azathioprine > 3 mg/kg/day, or any dose of cyclophosphamide, cyclosporine, or thalidomide;
* Have received leflunomide >20 mg/day in the 6 months prior to Study Day 0;
* Have received fluctuating doses of antimalarials, mycophenolate mofetil, methotrexate,leflunomide, or azathioprine within 28 days before randomization/entry or fluctuating doses of NSAIDs or oral corticosteroids within 14 days before randomization/entry;
* Treatment with any investigational drug therapy within 28 days before randomization/entry into the study, B cell-depleting therapies within 12 months before randomization/entry, or biologic therapies within 30 days or 5 half-lives of the biologic agent, whichever is longer,before randomization/entry into the study;
* In the investigator's opinion, evidence of clinically significant active infection, including ongoing, chronic infection, within 28 days before randomization/entry;
* A history of severe viral infection as judged by the investigators, including severe infections of either cytomegalovirus or the herpes family such as disseminated herpes, herpes encephalitis, ophthalmic herpes;
* Herpes zoster infection within 3 months before randomization/entry;
* Evidence of infection with hepatitis B or C virus, or HIV-1 or HIV-2, or active infection with hepatitis A, as determined by results of testing at screening;
* Vaccination with live attenuated viruses within 28 days before randomization/entry;
* Pregnancy (women, unless surgically sterile or at least 2 years post-menopausal, must have a negative serum pregnancy test within 28 days before receiving the study drug and a negative urine pregnancy test on Study Day 0 before receiving the study drug);
* Breastfeeding or lactating women;
* History of primary immunodeficiency;
* History of alcohol or drug abuse < 1 year prior to randomization/entry;
* History of cancer (except basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy > 1 year prior to randomization/entry);
* History of active TB infection;
* History of latent TB infection or newly positive TB skin test (reaction defined as ≥ 10 mm in diameter if not on systemic immunosuppressive medication or ≥ 5 mm if on systemic immunosuppressive medication) without completion of an appropriate course of treatment or with ongoing prophylactic therapy;
* Elective surgery planned from the time of screening through Study Day 196;
* At screening blood tests (within 28 days before randomization/entry), any of the following:

  * AST > 2 × upper limit of normal range (ULN), unless caused by SLE, as determined by the investigator,
  * ALT > 2 × ULN,unless caused by SLE, as determined by the investigator,
  * Creatinine > 4.0 mg/dL,
  * Neutrophils "1,500/ μL (< 1.5 × 109/L)"
  * Platelet count "Platelet count < 50,000/ μL (< 50 × 109/L)"
* History of any disease, evidence of any current disease (other than SLE), any finding upon physical examination, or any laboratory abnormality that, in the opinion of the investigator or medical monitor, may compromise the safety of the patient in the study or confound the analysis of the study; or
* Any employee of the research site who is involved with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2007-06; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of MEDI-545 will be assessed primarily by summarizing AEs and by assessing changes in viral cultures and titers. | Through Study Day 350.

SECONDARY OUTCOMES:
The secondary endpoints of this study are the PK and IM of multiple IV doses of MEDI-545. PK parameters, such as peak concentration. | Study day 350.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Greth, M.D., Study Director — MedImmune LLC
Locations (21):
- United States (16):
  - Research Site, Anniston, Alabama
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Clearwater, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Ocala, Florida
  - Research Site, Tampa, Florida
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Manhasset, New York
  - Research Site, New York, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Dallas, Texas
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, San Miguel de Tucumán
- Brazil (2):
  - Research Site, Curitiba, Paraná
  - Research Site, São Paulo
- Research Site, Santiago, Chile

REFERENCES:
- [Derived] Narwal R, Roskos LK, Robbie GJ. Population pharmacokinetics of sifalimumab, an investigational anti-interferon-alpha monoclonal antibody, in systemic lupus erythematosus. Clin Pharmacokinet. 2013 Nov;52(11):1017-27. doi: 10.1007/s40262-013-0085-2. PMID 23754736
- [Derived] Petri M, Wallace DJ, Spindler A, Chindalore V, Kalunian K, Mysler E, Neuwelt CM, Robbie G, White WI, Higgs BW, Yao Y, Wang L, Ethgen D, Greth W. Sifalimumab, a human anti-interferon-alpha monoclonal antibody, in systemic lupus erythematosus: a phase I randomized, controlled, dose-escalation study. Arthritis Rheum. 2013 Apr;65(4):1011-21. doi: 10.1002/art.37824. PMID 23400715